CLINICAL TRIAL: NCT05515718
Title: Effect of the Early Ultrasound-guided Femoral Nerve Block Performed by Emergency Physicians on Pre-operative Opioids Usage in Patients With Proximal Femoral Fractures: a Randomized Controlled Trial
Brief Title: Effect of the Early Ultrasound-guided Femoral Nerve Block Performed by Emergency Physicians on Pre-operative Opioids Usage in Patients With Proximal Femoral Fractures
Acronym: FORELEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORELEG
Record Dates: First submitted 2022-08-17; First posted 2022-08-25 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Femoral Fracture; Femoral Nerve Block
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard pain management (Active Comparator): Patients receive a standard analgesic treatment, in accordance with the latest international guidelines :
  * if pain EN is ≥ 3: Paracetamol 1g every 6 hours (age <75 years) or every 8 hours (# 75 years) and/or Tramadol 50 mg every 8 hours ;
  * and/or if verbal EN for pain is ≥ 7: intravenous morphine titration according to local protocol: 3 mg bolus if weight > 60 kg and age ≤ 80 years; Bolus of 2 mg if weight ≤ 60 kg and age ≤ 80 years ; Bolus of 1 mg if age>80 years, regardless of weight ; This bolus is repeated every 5 minutes until an EN≤ 3 is obtained.
  Interventions: Other: Standard pain management
- Femoral nerve block (Experimental): Patients receive a standard analgesic treatment, in accordance with the latest international guidelines 5,13,45: - if pain EN is ≥ 3:
  Paracetamol 1g every 6 hours (age <75 years) or every 8 hours (# 75 years) and/or Tramadol 50 mg every 8 hours; - and/or if verbal EN for pain is ≥ 7: intravenous morphine titration according to local protocol: 3 mg bolus if weight > 60 kg and age ≤ 80 years; Bolus of 2 mg if weight ≤ 60 kg and age ≤ 80 years ; Bolus of 1 mg if age>80 years, regardless of weight ; This bolus is repeated every 5 minutes until an EN≤ 3 is obtained.
  Interventions: Other: Femoral nerve block

INTERVENTIONS:
Other: Standard pain management — Patients undergo ultrasound-guided femoral nerve blockperformed by a trained emergency physician, under strict aseptic conditions After the femoral nerve block is performed, the patient is monitored and (BP, HR, SpO2, ECG) during 90 minutes.
  Arms: Standard pain management
Other: Femoral nerve block — Patients undergo ultrasound-guided femoral nerve blockperformed by a trained emergency physician under strict aseptic conditions, immediately after oral informed consent is obtained. After the femoral nerve block is performed, the patient is monitored and (BP, HR, SpO2, ECG) during 90 minutes.
  Arms: Femoral nerve block

SUMMARY:
In France, approximately 80,000 patients with a fracture of the upper extremity of the femur (femoral neck or trochanter) are admitted in the emergency department. This is a serious disease with a one-year mortality rate of 29% (i.e., 1 of 5 women and 1 of 3 men), and significant consequences on quality of life and autonomy. The morbidity of these fractures is closely related to the occurrence of altered mental status or delirium, before and after surgery. The diagnosis is based on clinical features and x-rays of the hip. These fractures are associated with severe level of pain, before and after the surgery. For emergency physicians, managing appropriately the pain is a common problem at the admission in the emergency room. Proper pain management is essential to ensure patients' comfort before surgery, but also to ensure their return to their previous functional and cognitive state after surgery. For patients, the goal of treatment is to regain walking as quickly as possible, while minimizing surgical and medical complications. However, severe pain induced by the fracture may lead to an acute altered mental status or delirium. In France, the latest guidelines about analgesia in emergency medicine reported that local anesthesia and loco-regional anesthesia (LRA) are useful and should be promoted in emergency medicine. In 2010, these guidelines proposed to perform LRA techniques such as iliofascial block more widely available. In 2016, the largest review of the literature on the use of regional nerve blocks for hip and femoral neck fractures in the emergency department [MEDLINE (1946-2014), EMBASE (1947-2014), CINAHL (1960-2014), and the Cochrane Central Register of Controlled Trials] indicated that the femoral nerve block was likely to be at least as effective as, if not superior to, standard analgesic practices for decreasing pain after ESF fracture.

The authors of the meta-analysis suggested the superiority of ultrasound guidance compared to anatomic techniques or use of neurostimulation for an adequate needle placement. Despite the increasing availability of ultrasound in the emergency department, recent literature supporting the efficacy of ultrasound-guided femoral nerve block, and the improvement of ultrasound skills in routine emergency medicine practice, the literature lacks of data about the effective duration of action, medication influence, and the occurrence of complications when an ultrasound-guided femoral nerve block is used by emergency physicians at the admission.

For patients with hip fractures, it is questioned if ultrasound-guided femoral block used early on admission in the emergency room is in more efficient than intravenous morphine titration in reducing opioid use before surgery? Our hypothesis is that early use of ultrasound-guided femoral nerve block in the emergency room decreases preoperative opioid use (intravenous and/or oral) in patients with proximal femoral fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient with a suspicion of proximal femoral fracture at the emergency triage, defined as direct traumatism on hip or fall associated with hip pain and/or clinostatism and/or lower extremity deformity with, typically, shortening of the externally rotated limb

  * Patient with a verbal numerical pain rating ≥ 7 on emergency triage
  * Patient with a diagnosis of ESF fracture made on x-rays in the emergency department
  * Patient with a normal lower extremity neurovascular examination
  * Anticipated preoperative delay of at least 3 hours
  * Patient affiliated to a health insurance plan
  * French-speaking patient
  * Patient or relative who has given free, informed and written consent

Exclusion Criteria:

* Patient with multiples trauma
* No surgical treatment decided by the orthopedic team
* Prior femoral nerve block performed during pre-hospital time
* Patient was not walking before the fracture
* Patient has received opioids prior to ED admission (by home caregivers or as part of usual treatment) or buprenorphine or nalbuphine
* Contraindications to opioids: acute respiratory failure, acute liver failure, epilepsy not controlled by treatment, allergy; documented severe intolerance to morphine
* Contraindications to loco-regional anesthesia: constitutional or acquired coagulation disorder (anticoagulant treatment, acute hepatic failure), skin infection or wound near to the potential injection site, acute failure of an underlying disease, allergy to Ropivacaine or chlorhexidine
* Patient already included in a type 1 interventional research protocol (RIPH1)
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Pregnant or breastfeeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Advantage of the echo-guided femoral nerve block | Day 2
  This outcome corresponds to the absolute difference in opioid utilization (intravenous or oral) during the first 48 hours after the emergency department triage between a group of patients receiving standard pain management (SPN) and a group of patients receiving femoral nerve block (FNB).

SECONDARY OUTCOMES:
Evaluate the benefit of early implementation of FNB on reducing time to pain control after emergency triage | Day 1
  This outcome corresponds to the difference between the groups the time (minutes) from emergency department triage to obtaining a verbal Numerical Pain Scale (NPS) ≤ 3 out of 10 at rest and in motion.
Evaluate the benefit of early implementation of FNB on reducing time to standing after surgery | Hours 72
  This outcome corresponds to the difference between groups in the time (hours) between surgery and standing autonomously.
Evaluate the benefit of early implementation of the FNB on reducing overall opioid use (IV and/or PO) during the hospital stay | Day 30
  This outcome corresponds to the difference between the groups in overall, intravenous or oral opioid use (mg) between emergency department triage and hospital discharge.
Evaluate the benefit of early implementation of FNB on reducing the occurrence of complications related to overall opioid use (intravenous and/or per os) | Day 30
  This outcome corresponds to the difference between the groups in the occurrence of opioid-related complications, overall, intravenous or per os during the hospital length of stay, and their description, between the two groups i.e.: urinary retention, acute altered mental mental status, delirium, dyspnea and/or desaturation ≤ 92%, nausea and/or vomiting and/ or constipation requiring treatment, a fall.
Evaluate the difficulty experienced by the emergency physician for the ultrasound location of the femoral nerve and for the injection technique of the local anesthetic | Day 1
  This outcome corresponds to the difficulty measured on a 5-point Likert scale for the ultrasound location of the femoral nerve and for the injection technique of the local anesthetic.
  A. About ultrasound guidance How would you rate the ease of locating the femoral nerve and injection site on ultrasound?
  1. Very easy
  2. Somewhat easy
  3. Undecided
  4. Somewhat difficult
  5. Very difficult B. About local anesthesia How would you rate the ease of the local anesthetic injection technique (needle location, aspiration test, local anesthetic injection)
  1. Very easy 2. Somewhat easy 3. Undecided 4. Somewhat difficult 5. Very difficult

CONTACTS AND LOCATIONS:
Overall Officials: Camille GERLIER, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Haleem S, Lutchman L, Mayahi R, Grice JE, Parker MJ. Mortality following hip fracture: trends and geographical variations over the last 40 years. Injury. 2008 Oct;39(10):1157-63. doi: 10.1016/j.injury.2008.03.022. Epub 2008 Jul 24. PMID 18653186
- [Background] Gerson LW, Emond JA, Camargo CA Jr. US emergency department visits for hip fracture, 1992-2000. Eur J Emerg Med. 2004 Dec;11(6):323-8. doi: 10.1097/00063110-200412000-00005. PMID 15542989
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Riddell M, Ospina M, Holroyd-Leduc JM. Use of Femoral Nerve Blocks to Manage Hip Fracture Pain among Older Adults in the Emergency Department: A Systematic Review. CJEM. 2016 Jul;18(4):245-52. doi: 10.1017/cem.2015.94. Epub 2015 Sep 10. PMID 26354332
- [Background] Mouzopoulos G, Vasiliadis G, Lasanianos N, Nikolaras G, Morakis E, Kaminaris M. Fascia iliaca block prophylaxis for hip fracture patients at risk for delirium: a randomized placebo-controlled study. J Orthop Traumatol. 2009 Sep;10(3):127-33. doi: 10.1007/s10195-009-0062-6. Epub 2009 Aug 19. PMID 19690943
- [Background] Holdgate A, Shepherd SA, Huckson S. Patterns of analgesia for fractured neck of femur in Australian emergency departments. Emerg Med Australas. 2010 Feb;22(1):3-8. doi: 10.1111/j.1742-6723.2009.01246.x. Epub 2009 Dec 14. PMID 20015246
- [Background] Foss NB, Kristensen BB, Bundgaard M, Bak M, Heiring C, Virkelyst C, Hougaard S, Kehlet H. Fascia iliaca compartment blockade for acute pain control in hip fracture patients: a randomized, placebo-controlled trial. Anesthesiology. 2007 Apr;106(4):773-8. doi: 10.1097/01.anes.0000264764.56544.d2. PMID 17413915
- [Background] Beaudoin FL, Haran JP, Liebmann O. A comparison of ultrasound-guided three-in-one femoral nerve block versus parenteral opioids alone for analgesia in emergency department patients with hip fractures: a randomized controlled trial. Acad Emerg Med. 2013 Jun;20(6):584-91. doi: 10.1111/acem.12154. PMID 23758305
- [Result] Gerlier C, Mijahed R, Fels A, Bekka S, Courseau R, Singh AL, Ganansia O, Chatellier G. Effect of early ultrasound-guided femoral nerve block on preoperative opioid consumption in emergency patients with hip fracture: a randomized trial. Eur J Emerg Med. 2024 Feb 1;31(1):18-28. doi: 10.1097/MEJ.0000000000001075. Epub 2023 Aug 24. PMID 37650732
- See also: Les modalités de prise en charge des fractures du col du fémur en France de 1998 à 2009 — https://drees.solidarites-sante.gouv.fr/publications/etudes-et-resultats/les-modalites-de-prise-en-charge-des-fractures-du-col-du-femur-0